CLINICAL TRIAL: NCT05394051
Title: Improving the Psychological Well-being and Burnout Due to the COVID-19 Pandemic in the Northwestern Medicine (NM) Healthcare Worker SARS-CoV-2 Cohort (Severe Acute Respiratory Syndrome - Coronavirus 2)
Brief Title: Psychological Well-being and Burnout in Healthcare Workers During the COVID-19 (Coronavirus Disease 2019) Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Charlesnika Evans, Professor, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00212515
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Burnout; Burnout, Professional; Work-related Illness; Work-Related Stress; SARS-CoV-2 Infection
Keywords: healthcare worker; psychological wellbeing; pandemic
MeSH Terms: conditions — COVID-19; Burnout, Psychological; Burnout, Professional; Occupational Stress

STUDY DESIGN:
Intervention Model Description: This is a single group randomized trial. After baseline measures of burnout, well-being, and health behaviors are obtained, participants will be recruited for participation in the Positive Affect Regulation sKills (PARK) intervention from the NM HCW SARS-CoV-2 Cohort via direct email. Interested individuals will be provided with the URL (Uniform Resource Locator) to complete eligibility screening via REDCap. All HCWs will be eligible to participate unless they have already been identified as a participant in a previous PARK trial. Once they agree to enroll, they will be randomized to participate in the intervention (PARK) or the 'wait list control' arm (No PARK, but offered at the end of follow-up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARK Now (Experimental): 6-Week Self-Guided Program: PARK Positive Emotion Skills: The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access. A week will consist of 1-2 days of didactic material and 5-6 days of real-life skills practice and reporting. The maximum amount of time engaged in the PARK program for any participant is 5 hours over the 6-week period, plus completion of the REDCap surveys assessments (burnout, well-being, health behaviors). The intervention will focus on developing the following skills that will be supplemented by home practice: (1) positive events, capitalizing, gratitude; (2) mindfulness; (3) positive reappraisal; (4) personal strength and achievable goals; (5) and self-compassion.
  PARK is delivered through the BrightOutcome online platform.
  Interventions: Behavioral: Positive Affect Regulation sKills (PARK)
- Wait List Control-PARK Later (No Intervention): Wait list controls will be assessed at similar time intervals and will be offered PARK at end of follow-up.

INTERVENTIONS:
Behavioral: Positive Affect Regulation sKills (PARK) — The goal of the PARK program is to reduce feelings of anxiety, depression, and social isolation, as well as increase well-being and a sense of meaning and purpose through the practice of positive emotion skills via a self-guided online platform.
  The total time involved from the beginning to the end of the intervention portion of the study is approximately 6 months (includes 6-week PARK course, baseline and follow-up assessments. Wait list controls will be assessed at similar time intervals and will be offered PARK at end of follow-up.
  Other Names: PARK
  Arms: PARK Now

SUMMARY:
Healthcare systems around the world have faced tremendous stress because of the COVID-19 pandemic. Healthcare workers (HCWs) (ie. physicians, nurses, and support staff), who serve as the foundation of the healthcare system, report high levels of psychological stress and burnout, which will likely worsen as the pandemic continues. The consequences of stress and burnout can reduce quality of life for providers and lead to adverse health behaviors (poor dietary choices, reduced physical activity, increased alcohol intake, increases in weight etc.) among HCWs. In addition, burnout can have dire consequences on healthcare delivery effectiveness including poor quality of care and significant cost implications due to medical errors and HCW absenteeism and turnover. In fact, annual estimates of burn-out related turnover range from $7,600 per physician to >$16,000 per nurse. However, programs focused on reducing burnout in HCWs have the potential to reduce costs to the healthcare system by $5,000 per HCW per year. Maintaining and recovering psychological and behavioral well-being is essential to ensuring we have a workforce that is resilient to acute and ongoing stressors such as the COVID-19 pandemic, ensuring that they are capable of providing the highest level of quality and compassionate care to patients. In this project, we will strengthen the resiliency of the Northwestern Medicine (NM) healthcare system by implementing an online psychological well-being intervention (PARK). We will assess HCW willingness to engage in PARK, which has been shown in other populations experiencing stress (e.g. dementia caregivers, general public coping with COVID-19) to be effective. We will also assess if the PARK is effective in reducing stress and associated-burnout, absenteeism, and intentions to leave the workforce in a subset of 750 persons who have been participating in a study of HCWs at NM since Spring 2020. In the entire cohort, we will measure the psychological well-being, levels of burnout, health behaviors, absenteeism, and plans to leave the workforce at three time periods: the start, middle, and end of the study period and assess whether they differ by HCW characteristics including gender, race, and role in health care. Results from this study will provide much-needed information: 1) about the current state of psychological well-being and burnout among NM HCWs, now over 1 ½ years into the pandemic; 2) on the role of an online wellness intervention to improve well-being during a protracted pandemic; and 3) about the contribution of PARK to reduce burnout, HCW absenteeism and turnover, and potential impacts on costs. PARK has the potential to have a significant impact on not only NM HCWs but also to be generalizable to other healthcare organizations for addressing burnout and to contribute to lessons learned on how to support HCWs responding to future pandemics; ensuring resiliency in the healthcare delivery system. In addition, we will work with our already engaged stakeholder committee to ensure results can provide actionable policy and fiscal insights. Future opportunities will include collaboration with other healthcare systems to expand roll-out of the successful PARK intervention.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had a catastrophic impact on the world, resulting in the death of millions of people. It has placed an especially immense burden on healthcare workers (HCWs) who report damaged psychological well-being. Recent evidence suggests the psychological impact is worsening as the pandemic persists. The objective of this project is to assess and intervene to improve the psychological well-being among HCWs who have been active throughout the ongoing pandemic response. We will evaluate the acceptability, feasibility and early effectiveness of an online psychosocial wellness intervention designed to reduce burnout and promote psychological wellness among HCWs and describe workplace and personal characteristics associated with stress and burnout.

Aim 1: Assess the psychological well-being (depression, anxiety, positive affect, meaning and purpose) and burnout in an existing cohort of 3,569 HCWs working at Northwestern Medicine (NM) during the COVID-19 pandemic using self-report questionnaires.

Hypothesis 1: Higher burnout scores and evidence of poor psychological well-being (high depression, and anxiety and low positive affect and meaning and purpose) will be observed in patient-facing HCWs than in administrators.

Aim 2: Explore the associations of psychological well-being and burnout scores with health and cardio-metabolic behaviors (i.e., sleep, physical activity) and health-related absenteeism.

Hypothesis 2: Higher levels of emotional well-being will be associated with healthy behaviors.

Aim 3: Evaluate the acceptability, feasibility, and effectiveness of the evidence-based Positive Affect Regulation sKills (PARK) intervention to improve psychological well-being and reduce burnout among HCWs in a randomized control trial (RCT) with a wait list control.

Hypothesis 3.1: Participants will find PARK acceptable and feasible.

Hypothesis 3.2: Compared to control participants, those who have access to the PARK intervention will show improvements in psychological well-being and burnout.

Long-term impact: Our study will provide the foundation for a future randomized trial to determine the effect of PARK on psychological well-being, burnout, and downstream health behaviors and health outcomes among HCWs coping with significant stress. The results of this study may be used to implement programs like PARK to strengthen the health care delivery system and provide needed support to HCWs as they continue to respond to this pandemic and prepare for future shocks to the healthcare system in Chicago and across the US.

b. Significance and contribution

Psychological stress and burnout are an ongoing significant threat to HCW well-being and to the health systems ability to continue to both respond to the pandemic and deliver quality, people centered care. Stress and burnout among HCWs have been linked to diminished quality of patient care, including lower patient satisfaction with care and increased likelihood of medical errors and adverse health behaviors in HCWs. Stress is the perception that the demands of a situation outweigh resources for coping with those demands. When stress is ongoing, as it has been during the pandemic, it can lead to burnout. The construct of burnout, developed in studies of human-services workers, is characterized by emotional exhaustion (feeling emotionally drained by contact with patients), depersonalization (extreme detachment from patients), and lack of personal accomplishment (feelings of incompetence and lack of job success).

This challenge of HCW stress and burnout preexisted the COVID-19 pandemic. An Agency for Healthcare Research and Quality (AHRQ) study found that over half of primary care physicians felt stressed because of time pressures and other work conditions. In a 2015 survey, the AMA (American Medical Association) estimated rates of burnout at 40% among physicians in the US. The presence of stress and burnout has been further intensified by COVID-19. The COVID-19 pandemic has had a significant impact on the health care workforce in the United States (US), where there have been 567,599 cases and 1,821 deaths from COVID-19 in HCWs as of October 1, 2021. For frontline caregivers, who have witnessed an even larger number of deaths in the US and around the world, the psychological toll of the pandemic has been substantial. During the first year of the pandemic, 30-63% of HCWs reported stress depending on the setting, with the highest rates among nurses. In fact, a Society of Critical Care Medicine survey found that self-reported stress scores nearly tripled during the COVID-19 pandemic and included high rates in the 3 main areas of burnout (chronic exhaustion, cynicism and perceived ineffectiveness). Of course HCWs simultaneously faced other life stressors related to the pandemic, such as family and other caregiver responsibilities (e.g. illness and death in their own networks, economic strains) as well as fear of transmission to their family and friends due to workplace exposures. This dual toll of workplace and household stressors has resulted in increased rates of burnout, resulting in absenteeism and loss of people from the health care field when they are needed most.

The challenges of stress and burnout need to be addressed for the COVID-19 pandemic and beyond to address the current crisis and ready the workforce for the next health system shock by broader system changes around work practices (that go beyond this project) but also by increasing individual resiliency through positive affect wellness interventions. We propose to study the levels of stress and burnout and associations with health behaviors and health-related absenteeism in an existing longitudinal cohort of 3,569 NM HCWs comprised of frontline providers and support and administrative staff. We will also test the acceptability, feasibility, uptake and early effectiveness of an adapted on-line evidence-based intervention (PARK) to improve psychological wellbeing and levels of job burnout among this group. PARK was adapted by Dr. Moskowitz from a previously validated wellness intervention found to improve depression, positive emotion, and other aspects of psychological well-being across a range of populations, but not HCWs. Results from this study will: 1) document psychological well-being, health and cardio-metabolic behaviors, and absenteeism in the entire cohort; 2) assess the feasibility of an intervention, previously shown to be efficacious in other populations; and 3) explore the effectiveness of the intervention by comparing psychological well-being and burnout in those assigned to the intervention compared to those in a waitlist control condition. We expect that PARK will improve overall stress, burnout, and well-being in NM HCWs.

ELIGIBILITY:
Inclusion Criteria:

* Northwestern Medicine Healthcare worker >18 years old
* Participants will be eligible if they are a participant in the NM HCW Serology Study and they provide electronic informed consent to participate.
* Pregnant women and all employees of Northwestern Medicine are eligible for study.

Exclusion Criteria:

* If the participant no longer works for Northwestern Medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Psychological well-being | Survey will be sent out at baseline
  Assess the psychological well-being (depression, anxiety, positive affect, meaning and purpose) and burnout in an existing cohort of 3,569 HCWs working at Northwestern Medicine (NM) during the COVID-19 pandemic using self-report questionnaires.
  Psychological well-being will be measured using the PROMIS (Patient-Reported Outcomes Measurement Information System)/NIH Toolbox. The PROMIS/NIH Toolbox measures of psychosocial well-being will be used to measure psychological well-being using a Computer Adaptive Test (CAT) on anxiety, depression, social isolation, positive affect, and meaning and purpose.
  Approach: Participants will complete a ~15-minute survey with questions on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as a baseline assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up assessment given to the trial participants.
Psychological well-being at 3 months | Survey will be sent out at 3 months
  Assess the psychological well-being (depression, anxiety, positive affect, meaning and purpose) and burnout in an existing cohort of 3,569 HCWs working at Northwestern Medicine (NM) during the COVID-19 pandemic using self-report questionnaires.
  Psychological well-being will be measured using the PROMIS/NIH Toolbox. The PROMIS/NIH Toolbox measures of psychosocial well-being will be used to measure psychological well-being using a Computer Adaptive Test (CAT) on anxiety, depression, social isolation, positive affect, and meaning and purpose.
  Approach: Participants will complete a ~15-minute survey with questions on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as an updated assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up assessment given to the trial participants.
Burnout | Survey will be sent out at baseline
  Assess the psychological well-being (depression, anxiety, positive affect, meaning and purpose) and burnout in an existing cohort of 3,569 HCWs working at Northwestern Medicine (NM) during the COVID-19 pandemic using self-report questionnaires.
  Burnout will be measured using the Oldenburg Burnout Inventory (OLBI) which is a validated 16-item inventory which measures affective, physical, and cognitive aspects of burnout across positive and negative framed items of two core dimensions: exhaustion and disengagement (from work).
  Approach: Participants will complete a ~15-minute survey with questions on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as a baseline assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up assessment given to the trial participants.
Burnout at 3 months | Survey will be sent out at 3 months.
  Assess the psychological well-being (depression, anxiety, positive affect, meaning and purpose) and burnout in an existing cohort of 3,569 HCWs working at Northwestern Medicine (NM) during the COVID-19 pandemic using self-report questionnaires.
  Burnout will be measured using the Oldenburg Burnout Inventory (OLBI) which is a validated 16-item inventory which measures affective, physical, and cognitive aspects of burnout across positive and negative framed items of two core dimensions: exhaustion and disengagement (from work).
  Approach: Participants will complete a ~15-minute survey with questions on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as an updated assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up assessment given to the trial participants.

SECONDARY OUTCOMES:
Cardio-metabolic behaviors and health-related absenteeism | Survey will be sent out at baseline.
  Explore the associations of psychological well-being and burnout scores with health and cardio-metabolic behaviors (i.e., sleep, physical activity) and health-related absenteeism.
  Cardio-metabolic behaviors and absenteeism will be measured via the NIH PhenX (Phenotypes and eXposures) toolbox and CDC (Centers for Disease Control) measures. Physical activity will be assessed in MET (metabolic equivalent task) /minutes week, a continuous variable, sleep quality will be determined using a continuous score with higher values reflecting more sleep disturbances, alcohol will be drinks per week and dietary composition will be assessed.
  Approach: Participants complete a ~15-minute survey on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as a baseline assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up given to the trial participants.
Cardio-metabolic behaviors and health-related absenteeism at 3 months | Survey will be sent out at 3 months
  Explore the associations of psychological well-being and burnout scores with health and cardio-metabolic behaviors (i.e., sleep, physical activity) and health-related absenteeism.
  Cardio-metabolic behaviors and absenteeism will be measured via the NIH PhenX toolbox and CDC measures. Physical activity will be assessed in MET (metabolic equivalent task) /minutes week, a continuous variable, sleep quality will be determined using a continuous score with higher values reflecting more sleep disturbances, alcohol will be calculated as drinks per week and dietary composition will be assessed.
  Approach: Participants will complete a ~15-minute survey with questions on psychological well-being, burnout, health and cardio-metabolic behaviors, and absenteeism. These data will serve as an updated assessment on the current mental and physical health of HCWs. The cohort will also receive the same assessments at the last follow-up assessment given to the trial participants.

CONTACTS AND LOCATIONS:
Overall Officials: Charlesnika Evans, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Valdivia N, Hirschhorn LR, Vu TH, Dubois C, Moskowitz JT, Wilkins JT, Evans CT. Utilization of at-home tests for coronavirus disease 2019 (COVID-19) among healthcare workers in Chicago. Antimicrob Steward Healthc Epidemiol. 2024 Apr 24;4(1):e58. doi: 10.1017/ash.2024.17. eCollection 2024. PMID 38698942
- [Result] Wilkins JT, Hirschhorn LR, Gray EL, Wallia A, Carnethon M, Zembower TR, Ho J, DeYoung BJ, Zhu A, Rasmussen-Torvik LJ, Taiwo B, Evans CT. Serologic Status and SARS-CoV-2 Infection over 6 Months of Follow Up in Healthcare Workers in Chicago: A Cohort Study. Infect Control Hosp Epidemiol. 2022 Sep;43(9):1207-1215. doi: 10.1017/ice.2021.367. Epub 2021 Aug 9. PMID 34369331
- [Result] Wilkins JT, Gray EL, Wallia A, Hirschhorn LR, Zembower TR, Ho J, Kalume N, Agbo O, Zhu A, Rasmussen-Torvik LJ, Khan SS, Carnethon M, Huffman M, Evans CT. Seroprevalence and Correlates of SARS-CoV-2 Antibodies in Health Care Workers in Chicago. Open Forum Infect Dis. 2020 Dec 9;8(1):ofaa582. doi: 10.1093/ofid/ofaa582. eCollection 2021 Jan. PMID 33447642
- [Result] Evans CT, DeYoung BJ, Gray EL, Wallia A, Ho J, Carnethon M, Zembower TR, Hirschhorn LR, Wilkins JT. Coronavirus disease 2019 (COVID-19) vaccine intentions and uptake in a tertiary-care healthcare system: A longitudinal study. Infect Control Hosp Epidemiol. 2022 Dec;43(12):1806-1812. doi: 10.1017/ice.2021.523. Epub 2021 Dec 27. PMID 34955103
- [Result] Stone TD, Lee C, Bannon J, Vu TT, Hirschhorn LR, Wilkins JT, Evans CT. Intentions for uptake of the coronavirus disease 2019 (COVID-19) vaccine booster in healthcare workers. Infect Control Hosp Epidemiol. 2023 Apr;44(4):690-692. doi: 10.1017/ice.2022.307. Epub 2023 Mar 13. No abstract available. PMID 36912328
- [Result] Moskowitz JT, Jackson KL, Cummings P, Addington EL, Freedman ME, Bannon J, Lee C, Vu TH, Wallia A, Hirschhorn LR, Wilkins JT, Evans C. Feasibility, acceptability, and efficacy of a positive emotion regulation intervention to promote resilience for healthcare workers during the COVID-19 pandemic: A randomized controlled trial. PLoS One. 2024 Jun 24;19(6):e0305172. doi: 10.1371/journal.pone.0305172. eCollection 2024. PMID 38913665
- [Result] Bannon J, Evans CT, Freedman M, Lee C, Vu TH, Wallia A, Wilkins JT, Moskowitz JT, Hirschhorn LR. Psychological wellbeing and the association with burnout in a cohort of healthcare workers during the COVID-19 pandemic. Front Health Serv. 2022 Oct 25;2:994474. doi: 10.3389/frhs.2022.994474. eCollection 2022. PMID 36925776
- [Result] Lee C, Vu TT, Fuller JA, Freedman M, Bannon J, Wilkins JT, Moskowitz JT, Hirschhorn LR, Wallia A, Evans CT. The association of burnout with work absenteeism and the frequency of thoughts in leaving their job in a cohort of healthcare workers during the COVID-19 pandemic. Front Health Serv. 2023 Nov 29;3:1272285. doi: 10.3389/frhs.2023.1272285. eCollection 2023. PMID 38093812